CLINICAL TRIAL: NCT00837525
Title: Validity of Biodegradable Injectable Implant for the Treatment of External Nasal Valve Collapse.
Brief Title: Validity Study of a Nasal Valve Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nasoform, LLC (Industry)
Responsible Party: Iyad Saidi, Nasoform
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVB
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Nasal Valve Collapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: nasal valve implant — Injectable implantation of a biodegradable material for support of the Nasal valve.

SUMMARY:
The purpose of this study is to determine if an implant material can be injected to repair nasal valve collapse.

ELIGIBILITY:
Inclusion Criteria:

* Has nasal valve collapse

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Nasal obstruction symptom scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Iyad S Saidi, MD PhD, Principal Investigator — Metropolitan ENT and Facial Plastic Surgery
Locations (1):
- Metropolitan ENT and Facial Plastic Surgery, Alexandria, Virginia, United States